## **Study of Humidified Air to Improve Mucociliary Clearance (MCC) in COPD:**

## NCT03935932

Tim Corcoran, Ph.D., Frank Sciurba, M.D. Pulmonary, Allergy and Critical Care Medicine University of Pittsburgh

June 5, 2023

## **Statistical Analysis Plan:**

We will plot normalized retention vs. time and compare the percentage of deposited material cleared at t=90 min and up to 6 hours on the intervention days. Areas above the curve 90 min clearance curve will also be compared. We will calculate the central deposition percentage of the Tc-SC aerosol to ensure that Tc-SC aerosol delivery was similar on both testing days.

Statistical comparisons will be made using paired non-parametric statistics to compare the baseline clearance day to the Airvo clearance day (Wilcoxon Signed Rank).